CLINICAL TRIAL: NCT06671613
Title: Evaluating the Impact of Intermittent Fasting in Combination With Checkpoint Inhibitors in Patients With Non-small Cell Lung Cancer
Brief Title: Evaluating a Fasting-mimicking Diet in Combination With Immunotherapy in Patients With Non-small Cell Lung Cancer
Acronym: Stage IV NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Indiana University (Other); US Department of Veterans Affairs Cooperative Studies Program (Network); L-Nutra Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ONCB-014-24S; 14094145/CX002843 (Other Grant/Funding Number: VA Clinical Science Research & Development)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Stage IV NSCLC; NSCLC; Immunotherapy; Fasting Mimicking Diet
Keywords: PD1 inhibitors; Phase 2; Open Label; NSCLC; Fasting
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fasting | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, phase 2, randomized (partial crossover design) study evaluating the feasibility of FMD in stage IV NSCLC patients receiving single agent checkpoint inhibitors. Participants will be randomized 1:1 in blocks of 3. There is no blinding or stratification. Patients with high PDL1 NSCLC will be randomized to two arms: (Arm 1) 3 cycles of RD+PD1 inhibitors followed by 3 cycles of FMD+PD1 inhibitors or (Arm 2) 3 cycles of FMD+PD1 inhibitors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular Diet (Active Comparator): Patients will eat a RD with the first 3 cycles, then receive 3 cycles of FMD as they continue cycles 4-6.
  Interventions: Combination Product: Regular Diet Plus FMD
- FMD (Experimental): Plant based diet program.
  Interventions: Dietary Supplement: FMD; Combination Product: Regular Diet Plus FMD

INTERVENTIONS:
Dietary Supplement: FMD — Plant-based diet program
  Other Names: Xentigen
  Arms: FMD
Combination Product: Regular Diet Plus FMD — Patients will eat a RD with the first 3 cycles, then receive 3 cycles of FMD as they continue cycles 4-6
  Other Names: Regular Diet Plus Xentigen

SUMMARY:
The purpose of this study is to learn the effects of fasting on cancer cells while you get maintenance treatment.

DETAILED DESCRIPTION:
Cancer cells use an increased supply of glucose to make energy and do not have protection against fasting that normal cells do. Because of this, researchers would like to study how fasting may help immunotherapy target cancer cells. Initial studies suggest that fasting may decrease the side effects of immunotherapy and increase the chances of your cancer responding to the immunotherapy. Patient populations will have non-small cell lung cancer in which pembrolizumab have been recommended to treat the cancer as part of standard care

ELIGIBILITY:
Inclusion Criteria:

* 18 years at the time of informed consent
* Ability to provide written informed consent and HIPAA authorization.
* Eastern cooperative group (ECOG) performance status of 0 to 2
* Newly diagnosed histologically or cytologically confirmed stage IV Non-Small Cell Lung Cancer (NSCLC). Patients with locally advanced NSCLC that are not candidates for definitive therapy but are candidates for trial are allowed per investigator discretion.
* BMI 19 kg/m2
* Patients should be enrolled prior to starting standard of care immunotherapy for the treatment of stage IV NSCLC. Patients should be on PD (L)1 inhibitor alone (i.e., with PD-L1 expression 50%) in the metastatic setting. The investigators will allow single agent pembrolizumab only as the checkpoint inhibitor.
* Patients requiring palliative radiation or definitive radiation to an oligometastatic disease prior to the initiation of single agent checkpoint inhibitors are allowed once radiation has been completed and patients have recovered from toxicities.

Exclusion Criteria:

* Self-reported weight loss of > 10% in the 6 weeks prior to study entry
* History of symptomatic hypoglycemia or uncontrolled diabetes
* Prior therapies with inhibitors of insulin growth factor I(IGF-1) such as Linsitinib or Picropodophyllin
* Concurrent use of somatostatin
* Concurrent use of immunosuppressive medications including sirolimus, tacrolimus, mycophenolate mofetil, azathioprine, prednisone, dexamethasone, or cyclosporine
* Significant food allergies which would make the subject unable to consume the food provided.
* History or current evidence of any uncontrolled medical or psychiatric condition, therapy that may confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the participating subject as deemed by the treating investigator.
* Pregnant or lactating females are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of fasting mimicking diet intervention | Through study completion up to 2 years.
  Feasibility will be defined as the proportion of the patients who can finish the 3 cycles FMD without serious adverse events. The investigators define FMD as being a feasible intervention in NSCLC receiving checkpoint inhibitors if 70% of patients on study complete 3 cycles of FMD.
Compliance | Through study completion up to 2 years.
  Compliance will be measured by analysis of daily food diaries at the end of each FMD cycle.

SECONDARY OUTCOMES:
Immune Mediated Toxicities | Through study completion up to 2 years.
  Toxicities as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Overall response rate (ORR) | Through study completion up to 2 years.
  ORR defined as complete response (CR) + partial response (PR) per RECIST 1.1 criteria.
Disease control rate (DCR) | Through study completion up to 2 years.
  Defined as Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) per RECIST 1.1
  .
Progression Free Survival (PFS) | Through study completion up to 2 years.
  Defined as time from day 1 of starting on study to disease progression by RECIST 1.1 or death from any cause.
Functional Assessment of Cancer Therapy-Lung-(FACT-L) | Through study completion up to 2 years.
  A 36-item, questionnaire measured on a 5-point Likert scale with response options ranging from "not at all" to "very much." Total scores are summed in the range of 0 to 136. Higher scores indicate better QOL.
European Organization for the Research and Treatment of Cancer Quality of Life -(EORTC QLQ-C30) | Through study completion up to 2 years.
  A 30-item questionnaire measured on a 4-point response option ranging from ("not at all," to "very much"), except the global QoL scale which, has a 7-point response from ("very poor" to "excellent"). Scores range from 0-100, a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (4):
- United States (4):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No